CLINICAL TRIAL: NCT01393418
Title: EPO: A Renal Biomarker After Cardiac Surgery
Brief Title: Evaluating Erythropoietin as an Indicator for Possible Kidney Injury After Cardiac Surgery
Acronym: EPO
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Yasser Kouatli, Clinical Lecturer, University of Michigan
Other Study IDs: HUM41529
Record Dates: First submitted 2011-07-12; First posted 2011-07-13 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Erythropoietin; Acute Kidney Injury; Renal Biomarker
Keywords: Erythropoietin; Cardiac Surgery; Renal Biomarker; Acute Kidney Injury; Hypothermic Circulatory Arrest
MeSH Terms: conditions — Acute Kidney Injury | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects undergoing cardiac surgery
  Interventions: Other: Cardiac Surgery

INTERVENTIONS:
Other: Cardiac Surgery

SUMMARY:
The purpose of the study is to evaluate kidney biomarkers and determine if there is a correlation between Erythropoietin (EPO) levels and acute kidney injury after cardiac surgery. An early biomarker for kidney injury may be helpful in identifying, monitoring and managing patients at risk for kidney failure after cardiac surgery. To evaluate Erythropoietin's role as a predictor of poor renal function in the immediate post-bypass period we plan to compare EPO levels to Neutrophil gelatinase-associated lipocalin (NGAL).

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a serious complication after cardiac surgery and cardio-pulmonary bypass. AKI is associated with high mortality.

Erythropoietin, a hormone produced by the kidneys, will be evaluated as a potential biomarker of kidney injury. Neutrophil gelatinase-associated lipocalin (NGAL) has been studied as a biomarker of kidney injury. Early kidney injury detection has been long sought and NGAL has been shown to be a promising biomarker. A troponinlike biomarker of AKI that is easily measured and capable of both early detection and risk stratification would represent an advancement in our ability to differentiate acute kidney injury from failure.

Investigating EPO as a biomarker may prove to have increased predictive value in the clinical care of cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery with cardiopulmonary bypass with DHCA
* Normal renal function or renal insufficiency-serum creatinine less than 2.5 mg/dL
* Adult male and female patients 18 years and older

Exclusion Criteria:

* VADS
* Emergent cases
* Prolonged hypoxemia before, during or after bypass
* End stage renal disease
* Patients receive erythropoietin receptor agonists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac surgery patients.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Renal injury/Failure | 18 Hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yasser El Kouatli, MD, Principal Investigator — Department of Anesthesiology, University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No